CLINICAL TRIAL: NCT04132908
Title: Clinical-nutritional Trial to Evaluate the Effect of an Extract of Sclerocaya Birrea on the Glycemic Profile in Prediabetic Subjects
Brief Title: Clinical Trial to Evaluate the Effect of an Extract of Sclerocaya Birrea on Prediabetic Subjects
Acronym: PRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-0006
Record Dates: First submitted 2018-04-19; First posted 2019-10-21 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sclerocarya birrea (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement: nutraceutical
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: nutraceutical — Subjects will consume two capsules at breakfast and dinner for ten weeks.
  Arms: Sclerocarya birrea
Dietary Supplement: Placebo — Subjects will consume two capsules at breakfast and dinner for ten weeks.
  Arms: Placebo

SUMMARY:
It consists in the intake, during a period of 10 weeks, of a nutraceutical (natural extract of Sclerocarya birrea). It is a clinical trial, during which certain parameters of the glucidic metabolism will be measured analytically. Other secondary variables such as lipid profile, inflammatory markers, blood pressure, endothelial function and body composition will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years.
* Diagnosis of prediabetes according to the American Diabetes Association.

  * Altered fasting glucose (95-125 mg / dl).
  * Glucose intolerance (oral glucose tolerance test with glycemia at 2 hours between 140 - 199 mg / dl).
  * Hemoglobin glycated between 5.7 and 6.4%.
* Subjects with body mass index between 18-35 Kg / m2.
* Stable food habits: there is no gain or weight loss of more than 5 kg in the ten weeks.
* I do not consume foods rich in Screrocaria Birrea.

Exclusion Criteria:

* Subjects with a history of any type of liver or kidney pathology.
* Use of medications that may interfere with glucose metabolism.
* Consumption of alcohol greater than 20 g / day.
* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Participation in another clinical trial in the three months prior to the study
* Lack of will or inability to comply with clinical trial procedures.
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
endothelial function | The measurements of endothelial function are taken with an ultrasound on two different occasions. The measurements will be made at baseline and after ten weeks of product consumption. Up to 10 weeks
  Changes in the dilatation of the Humeral artery.
blood samples | It is performed in the laboratory with the ILAB 600 analyzer. Blood samples are analyzed on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product. Up to 10 weeks
  Changes in glycemic profile
Physical activity test | Quality of life measurements are taken with physical activity test on two different occasions. The measurements are made at the beginning and after ten weeks of consumption of the product. Up to 10 weeks
  Change in physical activity with the World Physical Activity Questionnaire (GPAQ)
nutritional record | The dietary intake will be controlled by a diary in which meals will be recorded for three days and on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product. Up to 10 weeks
  Potential changes in the dietary survey were controlled with a food diary
body composition | Body measurements are taken with a Tanita on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product. Up to 10 weeks
  Changes in body composition were measured with a TANITA
glucose tolerance test | The glucose measurements in venous blood are taken with a glucometer on three different occasions (1: at baseline before consumption of the product, 2: at five weeks and 3: ten weeks after ingestion of the layer product observe the changes) .
  Venous blood samples are taken from the finger at different times.
blood samples | It is performed in the laboratory with the ILAB 600 analyzer. Blood samples are analyzed on two different occasions. The measurements are made at the beginning and after eight weeks of consumption of the product. Up to 10 weeks
  Changes in lipidic profile:( total cholesterol, HDL and LDL) , it will be measured in mg/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No